CLINICAL TRIAL: NCT00526617
Title: A Phase I Study of ABT-888 in Combination With Temozolomide (TMZ) in Subjects With Non-Hematologic Malignancies (NHM) and Metastatic Melanoma (MM)
Brief Title: A Phase I Study of ABT-888 in Combination With Temozolomide in Cancer Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M06-862
Record Dates: First submitted 2007-09-05; First posted 2007-09-10 (Estimated); Last update posted 2017-11-21 (Actual); Status verified 2012-01

CONDITIONS: Non-hematologic Malignancies; Metastatic Melanoma; Breast Cancer; Ovarian Cancer; Primary Peritoneal Cancer; Fallopian Tube Cancer; Hepatocellular Carcinoma
Keywords: Solid Tumor; Melanoma; Breast cancer; Ovarian cancer; Primary peritoneal cancer; Fallopian tube cancer; Hepatocellular carcinoma; HCC; BRCA deficient; BRCA mutation; Temozolomide; Temodar; TMZ; ABT-888; PARP inhibitor
MeSH Terms: conditions — Melanoma; Breast Neoplasms; Ovarian Neoplasms; Fallopian Tube Neoplasms; Carcinoma, Hepatocellular | interventions — veliparib; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Open Label (Experimental): Within each dose level, subjects are treated with the same regimen/doses of ABT-888 and TMZ.
  Interventions: Drug: ABT-888; Drug: Temozolomide

INTERVENTIONS:
Drug: ABT-888 — Oral capsules
Drug: Temozolomide — Oral capsules
  Other Names: Temodar; TMZ

SUMMARY:
This Phase I clinical trial is studying the side effects and best dose of ABT-888 when given together with Temozolomide (chemotherapy) in treating patients with solid tumors, including metastatic melanoma (MM), BRCA deficient breast, ovarian, primary peritoneal, or fallopian tube cancer, and hepatocellular carcinoma (HCC).

DETAILED DESCRIPTION:
A Phase 1, multicenter, dose-escalation study evaluating the safety and tolerability of the PARP inhibitor ABT-888 in combination with Temozolomide (TMZ) in subjects with non-hematologic malignancies (NHM), including metastatic melanoma (MM), BRCA deficient breast, ovarian, primary peritoneal, or fallopian tube cancer, and hepatocellular carcinoma (HCC).

ELIGIBILITY:
Inclusion Criteria:

Dose escalation and expanded safety cohorts

* Evaluable disease, histologically confirmed malignancy (metastatic or unresectable) and standard curative measures or other therapy that may provide clinical benefit do not exist or are no longer effective
* ECOG Performance Score less than or equal to 2
* Adequate hematologic, renal and hepatic function
* Normal sodium, calcium and magnesium levels
* Voluntarily signed informed consent

Expanded Safety Cohorts Only

* Population:
* Metastatic melanoma (MM)
* Hepatocellular carcinoma (HCC) Child Pugh Category A and B classification only
* BRCA deficient tumor status*: advanced breast cancer (with soft tissue disease), or advanced ovarian cancer, or advanced primary peritoneal cancer, or advanced fallopian tube cancer*

  *Patients must have histologically or cytologically confirmed solid tumors with a positive genetic test result documenting BRCA 1 or BRCA 2 mutation status, to be considered eligible.
* Serial tumor biopsies: Required for all subjects enrolled in one of the Expanded Low Dose Safety Cohorts.

Exclusion Criteria:

Dose Escalation and Expanded Safety Cohorts

* Known central nervous system (CNS) metastases or CNS primary cancer.
* Previous or current malignancies at other sites, except: adequately treated in situ carcinoma of cervix uteri; basal/squamous cell carcinoma of skin; previous malignancy considered cured.
* Previous history or current seizure disorder.
* Clinically significant and uncontrolled major medical condition(s) or any medical condition that places the subject at an unacceptably high risk for toxicities.
* Transplant recipients and patients receiving combination anti-retroviral therapy for HIV due to the use of immunosuppressant therapies.
* Lactating or pregnant female.
* Chemotherapy, immunotherapy, radiotherapy, biologic or any investigational therapy will not be allowed within either 4 weeks, or 5 half lives of a targeted therapy prior to study drug administration (Study Day 1).
* Prior therapy with regimens containing dacarbazine (DTIC) or TMZ is not permitted.
* Anti-cancer therapy is not permitted during the treatment portion of the study.
* Hormone therapy, bisphosphonates or LHRH-agonists for prostate cancer are permitted prior to and during the study.
* Significant adverse event or toxicity due to previous anti-cancer treatment that has not recovered to within one grade level (not to exceed Grade 2) of baseline.

Expanded Safety Cohorts Only:

* MM Only: Prior treatment with DNA damaging agents or cytotoxic chemotherapy including carboplatin, cisplatin, fotemustine, paclitaxel, vincristine, TMZ and DTIC.
* Prior therapy with biologic agents (including IL-2, interferon, bevacizumab, vaccines and immunostimulants) and signal transduction inhibitors (including sorafenib, erlotinib, sutent and elesclomol) are allowed.

Lower Dose Expanded Safety Cohorts Only

* Anti-coagulant restrictions for subjects that have tumor biopsies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2007-08; Primary Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose | Duration of Study
Safety and Tolerability | Duration of Study
Pharmacokinetic Profile | Duration of Study

CONTACTS AND LOCATIONS:
Overall Officials: Bhardwaj Desai, MD, Study Director — Abbott

REFERENCES:
- [Result] Nuthalapati S, Munasinghe W, Giranda V, Xiong H. Clinical Pharmacokinetics and Mass Balance of Veliparib in Combination with Temozolomide in Subjects with Nonhematologic Malignancies. Clin Pharmacokinet. 2018 Jan;57(1):51-58. doi: 10.1007/s40262-017-0547-z. PMID 28497258